CLINICAL TRIAL: NCT06470308
Title: Prescribing Outcomes of a General Practitioner-Targeted Deprescribing Educational Intervention in Older Adults With Polypharmacy: A Cluster Randomized Trial
Brief Title: Prescribing Outcomes of a GP-Targeted Deprescribing Educational Intervention: A Cluster Randomized Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Alexandros Paraskevopoulos, MD , PhD Candidate, University of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 93/12.06.2023
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Medication Overuse; Deprescriptions; Polypharmacy; Frailty Syndrome
MeSH Terms: conditions — Prescription Drug Overuse; Frailty | interventions — Medication Review; Deprescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): An educational intervention and training in deprescribing algorithms and deprescribing tools ( Beers Criteria) will be provided to the general practitioners caring for the patients selected in the intervention arm.
  Interventions: Other: Medication Reviews and Deprescribing
- Control Arm (No Intervention): No educational intervention will be provided to the general practitioners of the selected patients.

INTERVENTIONS:
Other: Medication Reviews and Deprescribing — General Practitioners will be given training and education in deprescribing algorithms and the conduction of medication reviews with the use of validated deprescribing tools such as the Beers Criteria.
  Arms: Intervention Arm

SUMMARY:
Polypharmacy is a common and growing public health concern across healthcare settings worldwide and is associated with an increased risk of inappropriate prescribing and adverse drug events. Deprescribing-defined as the supervised withdrawal of potentially inappropriate medications using structured tools and clinical judgment-has been proposed as a strategy to improve prescribing safety. In Greece, formal initiatives and evidence evaluating deprescribing interventions in primary care remain limited.

This study is a cluster randomized controlled trial evaluating the effect of an educational intervention for general practitioners (GPs) on prescribing safety in primary care. Participating GPs are randomized in an approximately 1:1 ratio to an intervention or control arm. GPs in the intervention arm receive structured education and training on medication review and deprescribing, including the use of validated deprescribing tools such as the Beers Criteria. GPs in the control arm provide usual care and do not receive any educational intervention.

Patients receiving care from participating GPs are recruited, and prescribing outcomes are assessed at the patient level. The primary outcome is change in prescription medications following the intervention, comparing patients cared for by GPs in the intervention arm versus those cared for by GPs in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling patients
* Age ≥ 65 years
* Receive at least 5 medication ( polypharmacy )

Exclusion Criteria:

* hospitalized or patients living in nursing home
* Incapable of giving written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Potentially Inappropriate Medication | 1 years
  Determine if there is reduction in potentially Inappropriate medication after a deprescribing education intervention
Number of medications | 1 year
  Determine if there is reduction in number of medications after a deprescribing education intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ioanna Tsiligianni, MD, PhD, Study Chair — Associate Professor in General Practice and Public Health, Department of Social Medicine, University of Crete
Locations (1):
- Primary Care Facilities, Heraklion, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No
All the data that will be collected, will be retained only during the period needed for the aims of this research. Technical and organizational measures will be taken in order to minimize potential loss, destruction or corruption of the data.After the completion of the thesis , all the data will be destroyed.